CLINICAL TRIAL: NCT01268475
Title: Impact of Pulmonary Resection on Exercise Capacity in Patients With Bronchiectasis
Brief Title: Exercise Capacity in Bronchiectasis Resection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Instituto do Coração HCFMUSP (Dr. Ricardo Mingarini Terra, MD, PhD), Instituto do Coração HCFMUSP
Other Study IDs: CAPPesq 0671/10
Record Dates: First submitted 2010-11-18; First posted 2010-12-30 (Estimated); Last update posted 2010-12-30 (Estimated); Status verified 2010-11

CONDITIONS: Bronchiectasis
Keywords: Bronchiectasis; Quality of Life; Respiratory Function Tests; Exercise Test
MeSH Terms: conditions — Bronchiectasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Bronchiectasis can be defined as an abnormal and irreversible dilatation of the bronchial tree due to repeated cycles of inflammation and infection, resulting in progressive loss of lung function. The surgical treatment by pulmonary resection or even lung transplantation is indicated in cases of bronchiectasis primary nonresponsive to appropriate medical treatment, or when associated with serious complications. There are few literature data on the influence of bronchiectasis in exercise capacity, quality of life and functional capacity, and the impact of lung resection in patients with this diagnosis. The primary objective of this study is to evaluate prospectively the impact of lung resection on exercise capacity in patients with clinical and radiological diagnosis of bronchiectasis. The secondary objective of this study is to evaluate the impact of lung resection on quality of life and lung function and to analyze the the presence of predictors of postoperative functional deterioration and the occurrence of complications.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and radiographic diagnosis of bronchiectasis;
* Lack of adequate response to clinical treatment after 1 year of follow-up and / or presence of disease complications;
* Agreement to participate of the study by signing of the Informed Consent Term

Exclusion Criteria:

* Comorbidities that prevent the patient to undergo general anesthesia;
* Musculoskeletal and/or psychomotor disability to perform pulmonary function tests and cardiopulmonary exercise tests;
* Inability to understand the quality of life questionnaires;
* Age over 90 years or less 18 years.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with clinical and radiological diagnosis of bronchiectasis recruited on Pulmonary Suppurative Disease Clinic of Thoracic Surgery Department
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2009-03

PRIMARY OUTCOMES:
Impact of Pulmonary Resection on Exercise Capacity | Change from Baseline in Exercise Capacity at 3 months and Change from Baseline in Exercise Capacity at 9 months
  Exercise Capacity will be assessed using Cardiopulmonary Exercise Test.

SECONDARY OUTCOMES:
Impact of Pulmonary Resection on Quality of Life. | Change from Baseline in Quality of Life at 3 months and Change from Baseline in Quality of Life at 9 months.
  Quality of life will be assessed using WHOQOL-Bref and SF-36 questionnaries.
Impact of Pulmonary Resection on Lung Function. | Change from Baseline in Lung Function at 3 months and Change from Baseline in Lung Function at 9 months.
  Lung Function will be assessed using Spirometry Test.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Sao Paulo Medical School - Heart Institute, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Mariani AW, Vallilo CC, de Albuquerque ALP, Salge JM, Augusto MC, Suesada MM, Pego-Fernandes PM, Terra RM. Preoperative evaluation for lung resection in patients with bronchiectasis: should we rely on standard lung function evaluation? Eur J Cardiothorac Surg. 2021 Jun 14;59(6):1272-1278. doi: 10.1093/ejcts/ezaa454. PMID 33491053